CLINICAL TRIAL: NCT03728803
Title: Inspiratory Muscle Training in Patients With Nemaline Myopathy
Brief Title: Inspiratory Muscle Training in Nemaline Myopathy
Acronym: NEMTRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: NL65214.091.18
Record Dates: First submitted 2018-10-15; First posted 2018-11-02 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2021-03

CONDITIONS: Nemaline Myopathy; Inspiratory Muscle Training
MeSH Terms: conditions — Myopathies, Nemaline

STUDY DESIGN:
Intervention Model Description: A controlled before-after trial of inspiratory muscle training will be performed in patients with nemaline myopathy with respiratory muscle weakness. The 2 sequentially tested conditions are sham IMT and active IMT. Patients are not blinded to the conditions, instead patients are instructed that two training methods are tested. First the effect of breathing technique with low resistance (sham IMT) and secondly with high resistance (active IMT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham inspiratory muscle training (Sham Comparator): Commercially available threshold IMT trainers (Threshold IMT, Philips Respironics) for inspiration will be used. For sham IMT the valve will be removed, creating a low resistance.
  The participants will perform the sham IMT twice a day during 15 minutes for a period of 8 weeks.
  Interventions: Device: Threshold IMT, Philips Respironics, Murrysville, PA, USA
- Active inspiratory muscle training (Active Comparator): Commercially available threshold IMT trainers (Threshold IMT, Philips Respironics) for inspiration will be used. After the sham IMT, the participants will perform an active inspiratory muscle training during 8 weeks with the same training schedule. The resistance will gradually be increased in the first couple of weeks until the intended resistance (30% of MIP) is reached.
  Interventions: Device: Threshold IMT, Philips Respironics, Murrysville, PA, USA

INTERVENTIONS:
Device: Threshold IMT, Philips Respironics, Murrysville, PA, USA — Active inspiratory muscle training (IMT) by the threshold IMT provides consistent and specific pressure for inspiratory muscle strength and endurance training, regardless of how quickly or slowly patients breathe. This device incorporates a flow-independent one-way valve to ensure consistent resistance and features an adjustable specific pressure setting (in cmH20) to be set. When patients inhale through the Threshold IMT, a spring-loaded valve provides a resistance that exercises respiratory muscles through conditioning.

SUMMARY:
Nemaline myopathy is a rare congenital myopathy. Respiratory failure is the main cause of death in these patients. The primary objective of this study is to determine the effect of a 8-week inspiratory muscle training program on respiratory muscle function in nemaline myopathy patients. The secondary objective is to determine respiratory muscle function in nemaline myopathy patients and its correlation with clinical severity and general neuromuscular function. The nemaline myopathy patients will be included in the first phase for a clinical characterization. From this phase patients will be selected for the second phase, which is a controlled before-after trial of inspiratory muscle training. The primary outcome is the change in maximal inspiratory pressure (MIP) after active inspiratory muscle training

DETAILED DESCRIPTION:
Rationale: Nemaline myopathy is a group of congenital, hereditary neuromuscular disorders with variable symptoms such as muscle weakness, swallowing dysfunction, and dysarthria. Respiratory failure is the main cause of death in nemaline myopathy and occurs even in ambulant patients who otherwise appear to be only mildly affected; respiratory muscle weakness may even be the presenting feature. Inspiratory muscle training has shown to increase inspiratory muscle strength in patients with other neuromuscular disorders. It is hypothesized that inspiratory muscle training improves respiratory muscle function in nemaline myopathy patients with respiratory muscle weakness.

Objective: The primary objective is to determine the effect of a 8-week inspiratory muscle training program on respiratory muscle function in nemaline myopathy patients. The secondary objective is to determine respiratory muscle function in nemaline myopathy patients and its correlation with clinical severity and general neuromuscular function.

Study design: The study consist of two phases. Phase 1: A screening phase with an open design from which patients will be selected for the second phase. Phase 2: A controlled before-after trial of inspiratory muscle training. The 2 conditions tested are sham IMT and active IMT.

Study population: Nemaline myopathy patients from the local neuromuscular database will be recruited. Furthermore, other centres in the Netherlands will be contacted to expand the database of nemaline myopathy patients. Phase 2 requires 23 patients.

Intervention: Active IMT consists of 15 minutes of IMT, twice a day, 5 days per week for 8 weeks, at a training workload of 30% of MIP using a resistive inspiratory muscle training device. Sham IMT consists of similar training regime using a resistive inspiratory muscle training device where the resistance has been removed.

Main study parameters/endpoints: The primary outcome parameter is the change in maximal inspiratory pressure (MIP) after active inspiratory muscle training.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The intervention of inspiratory muscle training is not associated with any risks, but can be challenging in patients with respiratory muscle weakness to perform. There will be three visits to the hospital in 16 weeks. The first visit has a maximal duration of 6 hours (including breaks) and the other two visits 1.5 hour. During these visits several tests and physical examinations will be performed. Some of the tests may cause some physical discomfort, but none of them carry any risk. Patients may benefit from participating in this study by developing improved respiratory muscle function as a result of the inspiratory muscle training.

ELIGIBILITY:
Inclusion Criteria:

* genetically-confirmed nemaline myopathy (mutations in one of the genes causing nemaline myopathy: TPM3, NEB, ACTA1, TPM2, TNNT1, KBTBD13, CFL2, KLHL40, KHLH41, LMOD3, MYPN, RYR1)
* informed consent from participant or legal representative
* age-range: between the age of 6-80 years

Exclusion Criteria:

* history of another condition that affects respiratory muscle strength or function (e.g. COPD)

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Change of maximal inspiratory pressure (cmH2O) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with handheld device

SECONDARY OUTCOMES:
Change of diaphragm thickness (mm) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with ultrasound
Change of diaphragm thickening (ratio) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with ultrasound
Change of diaphragm excursion (cm) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with ultrasound
Change of peak cough flow (L/s) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with handheld spirometry
Change of forced vital capacity (% predicted) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with handheld spirometry
Change of forced expiratory volume in the first second (% predicted) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with handheld spirometry
Change of peak expiratory flow (L/s) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with handheld spirometry
Change of (Slow) vital capacity (% predicted) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with handheld spirometry in sit and supine
Change of sniff nasal inspiratory pressure (cmH2O) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with handheld device
Change of maximal expiratory pressure (cmH2O) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Obtained with handheld device
Change of twitch mouth pressure (cmH2O) | Baseline, after 8 weeks sham IMT, after 8 weeks active IMT
  Measured after bilateral phrenic nerve stimulation
Maximal voluntary contraction (N) | Baseline
  Handgrip ergonometer
Rate of muscle relaxation (N/s) | Baseline
  Measured by transcranial magnetic stimulation
Motor Function Measure test | Baseline
  The items of the MFM are classified in 3 domains:
  D1: Standing and transfers (13 items, sub score range 0-39) D2: Axial and proximal motor function (12 items, sub score range 0-36) D3: Distal motor function (7 items, sub score range 0-21) Each item is scored on a 0-3 scale. Each sub score will be calculated as the percentage of total possible score achieved. Higher scores indicate a better outcome. The range of the total score is 0-96, again recalculated as the percentage of total possible score achieved.
6-minute walk test | Baseline
  This test assesses distance walked over 6 minutes as a submaximal test of aerobic capacity/endurance. The outcome is compared to the reference values.
Falls | 100-day period from baseline on
  The occurence of falls will be investigated retrospectively and prospectively during a 100-day period by questions composed by the investigators.
Mini-BESTest: Balance Evaluation Systems Test (Balance test for adults) | Baseline
  This test consists of several domains of balance and consequently of several sub scores:
  Anticipatory sub score 0-6 Reactive postural control 0-6 Sensory orientation sub score 0-6 Dynamic gait sub score 0-10
  The sub scores are added up to a total score with a range of 0-28. Higher values represent a better outcome.
Pediatric Balance Scale (Balance test for children) | Baseline
  This test consists of 14 item. The participant can score 0-4 on each item, with a maximum score of 56. Higher values represent a better outcome.
The RAND 36-Item Health Survey | Baseline
  This questionnaire addresses eight concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health.
  Scoring the RAND 36-Item Health Survey is a two-step process. First, precoded numeric values are recoded per the scoring key. All items are scored so that a high score defines a more favourable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are set at 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create the 8 scale scores. Hence, scale scores represent the average for all items in the scale that the respondent answered.
Measurement model for the pediatric quality of life inventory: PedsQL | Baseline
  This questionnaire consists of 8 items on physical functioning, 5 items on emotional functioning, 5 items on social functioning, and 5 items on school functioning. Each item is scored on a 0-4 scale. The items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate a better outcome. To create the Psychosocial Health Summary Score, the mean is computed as the sum of the items over the number of items answered in the Emotional, Social, and School Functioning Scales. The Physical Health Summary Score is the same as the Physical Functioning Scale Score. To create the Total Scale Score, the mean is computed as the sum of all the items over the number of items answered on all the Scales.

CONTACTS AND LOCATIONS:
Overall Officials: Baziel van Engelen, Prof. PhD, Study Director — Promotor
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided